CLINICAL TRIAL: NCT00028912
Title: Phase I Trial of Bortezomib (NSC 681239, IND#58443) and Carboplatin in Recurrent or Progressive Epithelial Ovarian Cancer or Primary Peritoneal Cancer
Brief Title: Bortezomib and Carboplatin in Treating Patients With Recurrent or Progressive Ovarian Epithelial, Primary Peritoneal, or Fallopian Tube Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000069146; MSKCC-01097; NCI-5326
Record Dates: First submitted 2002-01-04; First posted 2003-01-27 (Estimated); Last update posted 2011-04-26 (Estimated); Status verified 2004-04

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Primary Peritoneal Cavity Cancer
Keywords: recurrent ovarian epithelial cancer; primary peritoneal cavity cancer; fallopian tube cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Bortezomib; Carboplatin

INTERVENTIONS:
Drug: bortezomib
Drug: carboplatin

SUMMARY:
RATIONALE: Bortezomib may stop the growth of tumor cells by blocking the enzymes necessary for tumor cell growth. Drugs used in chemotherapy such as carboplatin use different ways to stop tumor cells from dividing so they stop growing or die. Bortezomib may help carboplatin kill more tumor cells by making tumor cells more sensitive to the drug.

PURPOSE: Phase I trial to study the effectiveness of combining bortezomib with carboplatin in treating patients who have recurrent or progressive ovarian epithelial, primary peritoneal, or fallopian tube cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of bortezomib in combination with carboplatin in patients with recurrent or progressive ovarian epithelial, primary peritoneal, or fallopian tube cancer.
* Determine the toxicity of this regimen in these patients.
* Determine the pharmacodynamics of this regimen in these patients by measurement of 20S proteasome inhibition in whole blood.
* Correlate toxicity with 20S proteasome inhibition in a whole blood assay in patients treated with this regimen.

OUTLINE: This is a dose-escalation study of bortezomib.

Patients receive carboplatin IV over 30 minutes on days 1 and 8 followed by 1 week of rest during the first course of treatment. Beginning with the second course, patients receive bortezomib IV on days 1, 4, 8, and 11 and carboplatin IV over 30 minutes on days 1 and 8. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of bortezomib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, 8 additional patients are accrued and treated at that dose.

PROJECTED ACCRUAL: A total of 3-32 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed ovarian epithelial, primary peritoneal, or fallopian tube cancer

  * Recurrent or progressive disease
* Received at least 1 prior platinum-based chemotherapy regimen containing carboplatin, cisplatin, or another organoplatinum compound for primary disease

  * May include high-dose therapy, consolidation, or extended therapy after surgical or non-surgical assessment
* No brain metastases or leptomeningeal involvement

PATIENT CHARACTERISTICS:

Age:

* Not specified

Performance status:

* Karnofsky 70-100%

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 1,000/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 8.0 g/dL

Hepatic:

* AST and ALT no greater than 2.5 times upper limit of normal
* Bilirubin no greater than 1.8 mg/dL

Renal:

* Creatinine no greater than 1.5 mg/dL

Cardiovascular:

* LVEF greater than 50% by radionuclide ventriculogram or two-dimensional echocardiogram
* No peripheral vascular disease requiring surgical management
* No prior myocardial infarction
* No congestive heart failure
* No orthostatic hypotension
* No acute ischemia or significant conduction abnormality (bifascicular block, defined as left anterior hemiblock with right bundle branch block, second or third degree AV blocks) as evidenced by electrocardiogram
* No prior cerebrovascular event

Other:

* No peripheral neuropathy grade 2 or greater
* No other serious medical or psychiatric illness
* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics
* No more than 2 prior regimens for recurrent disease, including 1 non-platinum containing regimen
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas and mitomycin) and recovered

Endocrine therapy:

* At least 1 week since prior hormonal therapy directed at primary tumor
* Concurrent hormone replacement therapy allowed

Radiotherapy:

* Not specified

Surgery:

* See Disease Characteristics
* At least 2 weeks since prior major surgery

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2001-11

CONTACTS AND LOCATIONS:
Overall Officials: Carol Aghajanian, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Result] Aghajanian C, Dizon DS, Sabbatini P, Raizer JJ, Dupont J, Spriggs DR. Phase I trial of bortezomib and carboplatin in recurrent ovarian or primary peritoneal cancer. J Clin Oncol. 2005 Sep 1;23(25):5943-9. doi: 10.1200/JCO.2005.16.006. PMID 16135465